CLINICAL TRIAL: NCT07143552
Title: A Prospective Case-Control Study of Vitamin D Status, Bone Metabolic Markers, and Overweight in Pediatric Low-Energy Fractures
Brief Title: Bone Outcomes, Obesity, Sunlight, and Trauma in Children
Acronym: BOOST
Status: Recruiting | Type: Observational
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Andrea Cosentino, Medical Doctor, Principal Investigator, Department of Orthopedics, Attending PhD, Paracelsus Medical University
Other Study IDs: prot. N. 0098306-BZ REG01
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Fractures; Hypovitaminosis D; Obesity and Overweight
Keywords: Vitamin D; Alkaline phosphatase; Calcium; Case-control; bmi; phosphate; Low-energy trauma
MeSH Terms: conditions — Vitamin D Deficiency; Obesity; Overweight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fracture group: Children aged 3-15 years with radiologically confirmed low-energy fractures.
- Control group: Children aged 3-15 years with low-energy trauma but no radiological evidence of fracture.

SUMMARY:
Prospective case-control study of children (3-15 years) after low-energy trauma. We compare serum bone metabolic markers (25OHD, PTH, ALP, calcium, phosphate), BMI/percentile, and dietary calcium intake between fracture and non-fracture presentations. Blood is collected within 7 days (non-fasting; samples on ice for PTH). Primary aim: association of ALP and calcium with fracture status; secondary aims: vitamin D status, BMI percentile, and a composite Bone Risk Score (≥3). Analyses: group comparisons, logistic regression, ROC.

DETAILED DESCRIPTION:
Low-energy fractures in children are a common cause of morbidity and may reflect underlying skeletal fragility. Emerging evidence suggests that hypovitaminosis D, obesity, and abnormal bone metabolism play important roles in fracture risk. However, the combined effect of these factors remains insufficiently studied, particularly in pediatric populations.

This study is designed as a prospective case-control investigation to explore the relationship between vitamin D status, bone metabolic markers, and obesity in children presenting with trauma. Children aged 3-15 years with low-energy trauma will be recruited and divided into two groups: those with radiologically confirmed fractures (cases) and those with similar trauma but without fractures (controls).

Baseline assessments include anthropometric measurements, dietary calcium intake through a food-frequency questionnaire, and laboratory evaluation of bone metabolism. Blood samples will be obtained within 7 days of the trauma and processed under standardized conditions to measure 25-hydroxyvitamin D (25OHD), parathyroid hormone (PTH), alkaline phosphatase (ALP), calcium, and phosphate. Samples are collected non-fasting and stored on ice to minimize variability in PTH measurement.

The primary outcome is the association of fracture occurrence with serum alkaline phosphatase (ALP) levels. Secondary outcomes include serum calcium, 25OHD concentration, a composite bone risk score, and body mass index (BMI) percentile. Outcomes are analyzed using descriptive statistics, group comparisons, and logistic regression to identify independent predictors of fracture risk.

The study aims to provide novel insights into the multifactorial etiology of pediatric fractures. By integrating metabolic, nutritional, and anthropometric data, the project seeks to establish a more comprehensive risk profile that can guide preventive strategies and inform clinical practice in pediatric bone health.

ELIGIBILITY:
Inclusion Criteria:

* 3-15 years;
* low-energy trauma;
* cases = radiographic fracture; controls = no fracture.

Exclusion Criteria:

* chronic renal/liver disease;
* primary hypo-/hyperparathyroidism;
* hypophosphatemic rickets;
* neuromuscular disorders;
* corticosteroids/bisphosphonates;
* unclear diagnosis/treatment.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children and adolescents aged 3 to 15 years presenting to emergency services after low-energy trauma. Eligible participants include those with radiologically confirmed fractures (case group) and those with comparable trauma without fractures (control group). All participants are otherwise healthy and free from chronic conditions or treatments that may influence bone metabolism.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Serum 25-hydroxyvitamin D (nmol/L) | within 7 days
  Blood level of vit D
BMI | at baseline
  Relation between BMI and Fracture

SECONDARY OUTCOMES:
Calcium, Phosphate, alkaline phosphatase | within 7 days from trauma
  Serum level of bone metabolism markers
bone risk score | at baseline
  proportion with score ≥3

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cosentino, MD, Principal Investigator — Franz Tappeiner Hospital; Paracelsus Medical University
Locations (2):
- Italy (2):
  - Kaiser Franz Joseph Hospital, Brixen, Bolzano
  - Franz Tappeiner Hospital, Meran, Bolzano

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gonzalez N, Nahmias J, Schubl S, Swentek L, Smith BR, Nguyen NT, Grigorian A. Obese adolescents have higher risk for severe lower extremity fractures after falling. Pediatr Surg Int. 2023 Jul 19;39(1):235. doi: 10.1007/s00383-023-05524-9. PMID 37466766
- [Background] Ergun T, Cansever M. Comparison of 25-OH vitamin D levels between children with upper and those with lower extremity fractures: A prospective case-control study. Acta Orthop Traumatol Turc. 2022 Mar;56(2):76-80. doi: 10.5152/j.aott.2022.21018. PMID 35416156
- [Background] Moore DM, O'Sullivan M, Kiely P, Noel J, O'Toole P, Kennedy J, Moore DP, Kelly P. Vitamin D levels in Irish children with fractures: A prospective case-control study with 5 year follow-up. Surgeon. 2022 Apr;20(2):71-77. doi: 10.1016/j.surge.2021.02.015. Epub 2021 Apr 24. PMID 33903053
- [Background] Yang G, Lee WYW, Hung ALH, Tang MF, Li X, Kong APS, Leung TF, Yung PSH, To KKW, Cheng JCY, Lam TP. Association of serum 25(OH)Vit-D levels with risk of pediatric fractures: a systematic review and meta-analysis. Osteoporos Int. 2021 Jul;32(7):1287-1300. doi: 10.1007/s00198-020-05814-1. Epub 2021 Mar 11. PMID 33704541
- [Background] Clark EM, Ness AR, Bishop NJ, Tobias JH. Association between bone mass and fractures in children: a prospective cohort study. J Bone Miner Res. 2006 Sep;21(9):1489-95. doi: 10.1359/jbmr.060601. PMID 16939408
- [Background] Munns CF, Shaw N, Kiely M, Specker BL, Thacher TD, Ozono K, Michigami T, Tiosano D, Mughal MZ, Makitie O, Ramos-Abad L, Ward L, DiMeglio LA, Atapattu N, Cassinelli H, Braegger C, Pettifor JM, Seth A, Idris HW, Bhatia V, Fu J, Goldberg G, Savendahl L, Khadgawat R, Pludowski P, Maddock J, Hypponen E, Oduwole A, Frew E, Aguiar M, Tulchinsky T, Butler G, Hogler W. Global Consensus Recommendations on Prevention and Management of Nutritional Rickets. J Clin Endocrinol Metab. 2016 Feb;101(2):394-415. doi: 10.1210/jc.2015-2175. Epub 2016 Jan 8. PMID 26745253